CLINICAL TRIAL: NCT03681691
Title: The Interaction Between Diabetes and Estradiol on Human Brain Metabolism in Postmenopausal Women
Acronym: E2T2D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00049740; R21AG054955 (NIH)
Record Dates: First submitted 2018-09-10; First posted 2018-09-24 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Type 2; Dementia
Keywords: women's health; estradiol; postmenopausal
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dementia | interventions — Ortho Evra

STUDY DESIGN:
Intervention Model Description: Primary Objective: The primary objective is to determine whether the effects of glucose and ketone body uptake to the brain in response to 8-week administration of transdermal 17β-estradiol differ in postmenopausal women with and without type 2 diabetes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post menopausal women with diabetes (Experimental): 8-week administration of transdermal 17β-estradiol (Climara) patch in postmenopausal women with type 2 diabetes
  Interventions: Drug: Estradiol patch
- Post menopausal women without diabetes (Experimental): 8-week administration of transdermal 17β-estradiol (Climara) patch in postmenopausal women without type 2 diabetes.
  Interventions: Drug: Estradiol patch

INTERVENTIONS:
Drug: Estradiol patch — transdermal 17β-estradiol patch
  Other Names: Climara patch

SUMMARY:
The primary aim of this study is to test whether type 2 diabetes interacts with estradiol on brain metabolism in vivo in humans. This will be accomplished by imaging brain metabolism using positron emission tomography before and after short-term administration of transdermal 17β-estradiol in 10 postmenopausal women with diabetes and 10 non-diabetic postmenopausal women.

DETAILED DESCRIPTION:
Epidemiological studies suggest there may be an interaction between type 2 diabetes and estrogen in postmenopausal women, such that diabetes may interact with estrogen levels over time to increase risk for dementia. The mechanism for this effect is now known. However, animal research suggests that it may occur through estrogen's effects on cellular metabolism of glucose and ketone bodies. The primary aim of this study is to test whether type 2 diabetes interacts with estradiol on brain metabolism in vivo in humans. This will be accomplished by imaging brain metabolism using positron emission tomography before and after short-term administration of transdermal 17β-estradiol in 10 postmenopausal women with diabetes and 10 non-diabetic postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female, postmenopausal, aged 60-80
4. Normal results on recommended healthcare screenings (e.g., mammogram, pap smear, colonoscopy)
5. BMI 20-35 kg/m2
6. No evidence of dementia or mild cognitive impairment (MoCA score >25)
7. Able to access reliable transportation to study and intervention visits

Exclusion Criteria:

1. Use of hormone replacement therapy within the past 3 months
2. History of renal, heart, liver, or neurological disease; head injury with loss of consciousness in the past 5 years; chronic pain, anxiety or depression
3. Presence of medical conditions that might contraindicate estrogen use (e.g., unexplained vaginal bleeding, history of reproductive tissue cancer, thrombosis)
4. Currently taking insulin, metformin, or any other drug or medication judged by the study physician to affect safety or research outcomes of interest
5. Involved in another research study
6. Contraindications for MRI or PET scanning
7. Current smoker

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hugenschmidt, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at the present time.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post Menopausal Women With Diabetes | Post Menopausal Women Without Diabetes
Started | 8 | 4
Completed | 6 | 3
Not Completed | 2 | 1
Not completed — COVID | 1 | 0
Not completed — prolonged bleeding | 1 | 0
Not completed — veins would not stay open during the PET scan. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post Menopausal Women With Diabetes | Post Menopausal Women Without Diabetes | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (6.1) | 70.3 (3.6) | 70.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)--Whole Brain
Description: Brain metabolism will be measured using PET tracers to examine brain glucose uptake (FDG PET). PET imaging data are co-registered to T1 structural MRI data to conduct region-of-interest based analyses. Absolute global and regional uptake of FDG will be quantified.
Time Frame: Baseline
Population: Non-Diabetes: n=2, technical error resulted in issues reconstructing PET images for one participant. Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: micromoles/min/100g tissue
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 2 | 6
micromoles/min/100g tissue | 12.28 (11.39) | 11.75 (12.42)

2. Primary Outcome: FDG PET--Whole Brain
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromoles/min/100g tissue
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 2 | 6
micromoles/min/100g tissue | 8.74 (2.59) | 6.87 (0.88)

3. Primary Outcome: Acetoacetate Uptake (AcAc) PET--Whole Brain
Description: Brain metabolism will be measured using PET tracers to examine brain ketone body (acetoacetate) uptake (AcAc). PET imaging data are co-registered to T1 structural MRI data to conduct region-of-interest based analyses. Absolute global and regional uptake of AcAc tracers will be quantified.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromoles/min/100g tissue
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 2 | 6
micromoles/min/100g tissue | 0.031 (0.009) | 0.024 (0.005)

4. Primary Outcome: AcAc PET--Whole Brain
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromoles/min/100g tissue
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 2 | 6
micromoles/min/100g tissue | 0.027 (0.003) | 0.028 (0.015)

5. Primary Outcome: Change in Uptake of Glucose and Ketone Bodies in Whole Brain and Alzheimer's Disease-related Regions of Interest.
Description: Brain metabolism will be measured using PET tracers to examine brain glucose uptake (FDG PET) and ketone body (acetoacetate) uptake (AcAc). PET imaging data are co-registered to T1 structural MRI data to conduct region-of-interest based analyses. Absolute global and regional uptake of FDG and AcAc tracers will be quantified, as well as uptake of AcAc relative to FDG to find potential regions of compensatory ketone use
Time Frame: Baseline and 8 weeks
Population: This outcome measure is actually many outcome measures. It was broken down into the other four primary outcome measures listed, so no no results will be listed here. Also, rather than "change in", results will be reported as mean/standard deviation in the other outcomes.
Arm/Group | Post Menopausal Women With Diabetes | Post Menopausal Women Without Diabetes
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Short-Term Memory Composite Score
Description: A composite memory score was created by averaging z-scores for CVLT delayed recall, BVRT delayed recall, and prospective memory. A composite executive function score was created by averaging digit span forwards total correct, digit span backwards total correct, and both verbal fluency scores. Summed z-score ranging from -2 to 2 where higher score indicates better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
z-score
  Baseline | 1.04 (0.31) | -0.52 (2.01)
  Week 8 | 1.56 (0.53) | -0.56 (2.04)

7. Secondary Outcome: Executive Function Composite Score
Description: The California Verbal Learning Test (CVLT) is a word list recall task that can be used to test immediate and delayed verbal memory. Free recall after the short delay (immediately after learning lists) and long delay (25 minutes) are reported. Summed z-score ranging from -2 to 2 where higher score indicates better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
z-score
  Baseline | 0.20 (1.36) | -0.10 (1.78)
  Week 8 | 1.66 (4.83) | 0.30 (5.78)

8. Secondary Outcome: California Verbal Learning Task (CVLT) Long Delay Free Recall
Description: The CVLT is a word list recall task that can be used to test immediate and delayed verbal memory. Free recall after long delay (25 minutes). The minimum score is 0. The maximum score is 16 and a higher score represents better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
score on a scale
  Baseline | 12.0 (4.36) | 10.83 (3.25)
  Week 8 | 12.67 (2.08) | 13.17 (2.14)

9. Secondary Outcome: CVLT Short Delay Free Recall
Description: The CVLT is a word list recall task that can be used to test immediate and delayed verbal memory. Short delay free recall is immediately after learning lists. The minimum score is 0. The maximum score is 16 and a higher score represents better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
score on a scale
  Baseline | 11.67 (2.08) | 10.00 (3.91)
  Week 8 | 12.33 (1.15) | 11.67 (3.93)

10. Secondary Outcome: Benton Visual Retention Task (BVRT) Total Score
Description: The BVRT tests figural memory by testing memory for a line drawing. The minimum score is 0. The scoring used is total correct, the maximum score is 10, and a higher score represents better performance. The total score is reported.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
score on a scale
  Baseline | 8.67 (0.58) | 6.5 (2.07)
  Week 8 | 9.33 (0.58) | 5.5 (2.51)

11. Secondary Outcome: Prospective Memory
Description: The Prospective Memory test is a test of everyday memory where participants are given instructions for 3 tasks that will occur later on during the testing session. The minimum score is 0. The maximum score is 12 points, a higher score represents better performance, and the total score is reported
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
score on a scale
  Baseline | 10.67 (1.53) | 5.83 (3.97)
  Week 8 | 10.0 (2.0) | 8.17 (1.72)

12. Secondary Outcome: Verbal Fluency (Letters)
Description: Participants were given a letter and asked to say aloud as many words as they could think of beginning with that letter. The three letters were F, A, and S, and the participant had one minute per letter to list words. The total score reported is the sum of the correct words generated for all three letters. Although there is no set maximum score, based on published data, it was anticipated that scores could range from 1 to no more than 120. A higher value reflects better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: number of correct words generated
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
number of correct words generated
  Baseline | 48.67 (16.50) | 42.67 (9.56)
  Week 8 | 46.33 (12.58) | 41.33 (7.66)

13. Secondary Outcome: Verbal Fluency Score (Fruits and Vegetables)
Description: Participants were given one minute to say aloud as many fruits as possible and one minute to list as many vegetables as possible. The total score reported is the sum of all correct fruits and vegetables listed. Although there is no set maximum score, it was anticipated that scores could range from 0 to no more than 60. A higher value reflects better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: number of correct fruits and vegetables
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
number of correct fruits and vegetables
  Baseline | 31.0 (4.36) | 28.67 (8.62)
  Week 8 | 32.67 (7.23) | 29.17 (8.28)

14. Secondary Outcome: Digit Span Forward Total Correct
Description: Participants listened to a sequence of two to nine numbers and were asked to repeat each sequence back to the tester in the same order the numbers were presented. The outcome measure reported here is the total number of correct responses (range of scores 0-9). Higher scores reflect better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
number of correct responses
  Baseline | 8.0 (0.0) | 7.5 (0.55)
  Week 8 | 7.67 (2.08) | 7.67 (2.07)

15. Secondary Outcome: Digit Span Backward Total Correct
Description: Participants listened to a sequence of two to nine numbers and were asked to repeat each sequence back to the tester in reverse order. The outcome measure reported here is the longest span of numbers recalled (range of scores 0-9). Higher scores reflect better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: span of numbers recalled
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
span of numbers recalled
  Baseline | 4.0 (1.73) | 4.67 (0.82)
  Week 8 | 6.0 (1.0) | 5.33 (2.07)

16. Secondary Outcome: Finger Tapping Score--Dominant Hand
Description: The Finger Tapping test assesses fine motor speed by asking participants to tap a button as many times as possible. Seven trials were administered. The highest and lowest scores were dropped, and the reported score is the average of the remaining 5 trials. Results for the dominant hand are reported here. There is no set maximum score. However, published averages for women in this age range suggest that a value over 57 would be highly unusual. A higher value (more taps) is better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: number of taps
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
number of taps
  Baseline | 40.47 (4.65) | 43.53 (6.45)
  Week 8 | 40.27 (2.25) | 44.07 (5.2)

17. Secondary Outcome: Finger Tapping Score--Non-Dominant Hand
Description: The Finger Tapping test assesses fine motor speed by asking participants to tap a button as many times as possible. Seven trials were administered. The highest and lowest scores were dropped, and the reported score is the average of the remaining 5 trials. Results for the non-dominant hand are reported here. There is no set maximum score. However, published averages for women in this age range suggest that a value over 57 would be highly unusual. A higher value (more taps) is better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: number of taps
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
number of taps
  Baseline | 39.4 (4.1) | 38.2 (5.6)
  Week 8 | 42.7 (3.5) | 41.7 (6.7)

18. Secondary Outcome: Card Rotations Test Score
Description: The Card Rotations Test is used to assess the ability to mentally rotate figures in space. The test has two parts, each of which last 3 minutes. During each part, the participant is given a sheet of paper with 10 simple geometric figures. Next to each figure is a row of 8 similar figures. Participants are asked to mark whether each of the figures in the row is the same or different than the first figure in the row. The score reported is the number of correct responses. The minimum score is 0. The maximum possible score is 160 and a higher score reflects better performance.
Time Frame: Baseline and Week 8
Population: Results only reported for subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
Number analyzed (Participants) | 3 | 6
score on a scale
  Baseline | 76.0 (35.59) | 90.67 (34.60)
  Week 8 | 89.33 (5.86) | 97.0 (28.71)

19. Secondary Outcome: Change in Short-term Memory and Executive Function Composite Scores.
Description: A battery of cognitive tasks will be administered before and after estrogen administration. Composite z-scores will be calculated by calculating a z-score for each cognitive task and summing z-scores from -5 (low) to 5 (high) for the tasks designated as short-term memory and executive function.Higher scores denotes better outcomes.
Time Frame: Baseline and 8 weeks
Population: This outcome should have been separated into many other outcomes. So we have separated out all the scores and results will be reported in the other separated memory and executive function score outcomes. No results will be reported in this outcome. Also, rather than "change in", results will be reported as mean/standard deviation in the other outcomes.
Arm/Group | Post Menopausal Women With Diabetes | Post Menopausal Women Without Diabetes
Number analyzed (Participants) | 0 | 0

20. Other Pre Specified Outcome: Regional Ratio of Ketone/Glucose Uptake
Time Frame: Baseline and Week 8
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Number of White Matter Hypertensities
Description: Attained from a T2-weighted FLAIR image, an indicator of small-vessel disease correlated with diabetes status and hypertension
Time Frame: Baseline and Week 8
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of Microbleeds
Description: Attained from a susceptibility-weighted image
Time Frame: Baseline and Week 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Post Menopausal Women Without Diabetes | Post Menopausal Women With Diabetes
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 2/4 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Menopausal Women Without Diabetes (N=4) | Post Menopausal Women With Diabetes (N=8)
Elevated Blood Pressure (Vascular disorders) | 1 (1) | 0 (0)
Started Period-Like Bleeding/Spotting (Reproductive system and breast disorders) | 1 (1) | 5 (6)
Breast Tenderness/Soreness (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Cramping (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Itching Around Drug Patch (Product Issues) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fall at Home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03681691/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03681691/ICF_000.pdf